CLINICAL TRIAL: NCT07392008
Title: PASO A PASO Pilot Study: Tailored Diabetes Prevention Program for Spanish-Speaking Communities Feasibility Study
Brief Title: PASO A PASO: Tailored Diabetes Prevention Program for Spanish-Speaking Communities Feasibility Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Margaret (Molly) B. Conroy, Professor and Chief, Division of General Internal Medicine, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00183257
Record Dates: First submitted 2026-01-07; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Pre Diabetic
Keywords: feasibility; Spanish-speaking populations; diabetes prevention adaptation
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Feasibility and pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-based organizations leaders and community members (Experimental): Paso a Paso is a 12-month program designed for H/L community members who are at high risk for T2D and want to lower their risk.
  Interventions: Behavioral: Paso a Paso

INTERVENTIONS:
Behavioral: Paso a Paso — Cultural components will include fostering a sense of belonging, collaboration, support, interaction, and respect. Program structure: Paso a Paso is designed to include weekly 90-minute in-person sessions over the first 4 months of the program, which will transition to monthly sessions over the final 8 months of the intervention. All sessions will include hands-on skill development, group and social activities, and addressing assets for diabetes prevention available in the community. Finally, the intervention also includes an online community forum to support ongoing social support and information provision.

SUMMARY:
The interdisciplinary and interprofessional community-academic partnership (CAP) has been working with Spanish-speaking H/L Salt Lake City residents and organization leaders to adapt the National Diabetes Prevention Program to meet the needs of this population. This next collaboration phase attempts to finalize the adapted diabetes prevention program, "Paso a Paso," and evaluate its feasibility and implementation strategies. The purpose of this pilot study is to inform the necessary modifications to the Paso a Paso diabetes prevention intervention, ensuring that the full-scale future intervention is both feasible and effective for the target community.

DETAILED DESCRIPTION:
Specific goals include:

1. Finalize the adapted "Paso a Paso" protocol and materials.
2. Train the first cohort of instructors for the program (10-15 potential instructors)
3. Test the feasibility of the intervention implementation with 30 community participants.
4. Gather feedback from participants, refine the intervention, and ensure that it resonates with community members, ultimately laying the foundation for a successful larger study.

ELIGIBILITY:
Inclusion Criteria: Native Spanish speakers, residents in the Wasatch Front Metropolitan area, adults aged >18 years old with a BMI of ≥ 25, and diabetes risk >1 based on the CDC Prediabetes Risk Test

Exclusion Criteria:

1. Bariatric surgery in the last 2 years or planned during the next year
2. Edematous state that interferes with body weight assessment (e.g., severe congestive heart failure, end-stage renal disease, or ascites)
3. Current or planned pregnancy in the next year
4. Current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Weight percent change | Baseline, 4-month, 12-month (exploratory)
  Will be measured in kilograms using a calibrated Tanita WB-100A scale.

SECONDARY OUTCOMES:
% HbA1c | Baseline, 4-month, 12-month (exploratory)
  HbA1c will be tested using Point-of-Care (POC) A1c testing, which will require a finger prick.

OTHER OUTCOMES:
Waist circumference | Baseline, 4-month, 12-month (exploratory)
  Will be measured in centimeters using Gulick tape and standard research protocols.
Physical activity | Baseline, 4-month, 12-month (exploratory)
  Attendance in PA sessions
Dietary intake | Baseline, 4-month, 12-month (exploratory)
  Mediterranean Diet Score
Engagement measures | Baseline, 4-month, 12-month (exploratory)
  Retention, engagement, attendance rate (%)
Feasibility, acceptability, and appropriateness surveys | Baseline, 4-month, 12-month (exploratory)
  Validated a 5-point Likert scale to evaluate if an intervention is appealing, fits the context, and can be implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Molly B Conroy, MD, MPH, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with qualified researchers upon reasonable request, following publication of the primary study results.
Supporting Information: Study Protocol
Time Frame: 01/2027-01/2028
Access Criteria: Access will be limited to investigators with demonstrated scientific merit and the capacity to securely manage human subjects data. Shared data will exclude direct identifiers and comply with IRB approvals and HIPAA requirements for data-sharing expectations.

REFERENCES:
- [Background] Wells R, Yates L, Morgan I, deRosset L, Cilenti D. Using the Wilder Collaboration Factors Inventory to Strengthen Collaborations for Improving Maternal and Child Health. Matern Child Health J. 2021;25(3):377-84. Epub 2020/11/29. doi: 10.1007/s10995-020-03091-2. PubMed PMID: 33247823; PMCID: PMC7956933.
- [Background] Ritchie ND, Sauder KA, Phimphasone-Brady P, Amura CR. Rethinking the National Diabetes Prevention Program for low-income whites. Diabetes care. 2018;41(4):e56-e7. doi: 10.2337/dc17-2230.
- [Background] Mattessich PW, Johnson KM. Collaboration: What Makes It Work: Turner Publishing Company; 2018.
- [Background] Ritchie ND, Christoe-Frazier L, McFann KK, Havranek EP, Pereira RI. Effect of the National Diabetes Prevention Program on weight loss for English- and Spanish-speaking Latinos. Am J Health Promot. 2017;32(3):812-5. doi: 10.1177/0890117117698623.
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. The New England journal of medicine. 2001;344(18):1343-50. Epub 2001/05/03. doi: 10.1056/nejm200105033441801. PubMed PMID: 11333990.
- [Background] The National Registry of Recognized Diabetes Prevention Programs 2024: Centers for Disease Control and Prevention; [cited 2024 March 24]. Available from: https://dprp.cdc.gov/Registry.
- [Background] Ritchie ND, Baucom KJ, Sauder KA. Current perspectives on the impact of the National Diabetes Prevention Program: building on successes and overcoming challenges. Diabetes Metab Syndr Obes. 2020;13:2949-57. doi: 10.2147/dmso.s218334.
- [Background] Diabetes Prevention Program Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes care. 2002;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PubMed PMID: 12453955; PMCID: PMC1282458.
- [Background] López L, Golden SH. A new era in understanding diabetes disparities among U.S. Latinos-all are not equal. Diabetes care. 2014;37(8):2081-3. doi: 10.2337/dc14-0923.
- [Background] National diabetes statistics report: Centers for Disease Control and Prevention; 2024 [updated May 5, 2024; cited 2024 June 30]. Available from: https://www.cdc.gov/diabetes/php/data-research/index.html#:~:text=Among%20the%20U.S.%20population%20overall,Table%201a%3B%20Table%201b).
- [Background] Alemán JO, Almandoz JP, Frias JP, Galindo RJ. Obesity among Latinx people in the United States: A review. Obesity. 2023;31(2):329-37. doi: 10.1002/oby.23638.
- [Background] Vespa J, Medina L, Armstrong D. Demographic turning points for the United States: population projections for 2020 to 2060: US Census Bureau; 2020 [updated February 2020; cited 2024 July 27]. Available from: https://www.census.gov/content/dam/Census/library/publications/2020/demo/p25-1144.pdf.
- [Background] Community Research Collaborative. (2021). In it together: Community-based research guidelines for communities and higher education. Salt Lake City, UT: University of Utah.